CLINICAL TRIAL: NCT00801853
Title: A Phase IIb Study to Investigate the Treatment-Sparing Effects of AEROVANT™ AER 001 Inhalation Powder in Asthma Patients Not Fully Controlled on Current Therapy
Brief Title: A Study of the Treatment-Sparing Effects of AEROVANT™ AER 001 Inhalation Powder in Asthma Patients, AEROTRIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerovance, Inc. (Industry)
Responsible Party: Babatunde Otulana, M.D., Aerovance, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PPD/2007/AER 001 DPI/2b
Record Dates: First submitted 2008-12-01; First posted 2008-12-04 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2009-11

CONDITIONS: Asthma
Keywords: asthma; allergy; atopy; atopic; wheeze
MeSH Terms: conditions — Asthma; Hypersensitivity; Respiratory Sounds | interventions — pitrakinra

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerovant 1 (Experimental): Aerovant 1mg bid
  Interventions: Drug: Aerovant
- Aerovant 2 (Experimental): Aerovant 3mg bid
  Interventions: Drug: Aerovant
- Aerovant 3 (Experimental): Aerovant 10mg bid
  Interventions: Drug: Aerovant
- Placebo Control (Placebo Comparator): Placebo Control
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Aerovant — Aerovant 1mg bid (dry powder)
  Other Names: AER 001 DPI, BAY 16-9996, pitrakinra
  Arms: Aerovant 1
Drug: Aerovant — Aerovant 3mg bid (dry powder)
  Other Names: AER 001 DPI, BAY 16-9996, pitrakinra
  Arms: Aerovant 2
Drug: Aerovant — Aerovant 10mg bid (dry powder)
  Other Names: AER 001 DPI, BAY 16-9996, pitrakinra
  Arms: Aerovant 3
Other: placebo — placebo control (dry powder)
  Arms: Placebo Control

SUMMARY:
A multi-center, Phase IIb, double-blind, randomized, placebo controlled, parallel-group, repeated-dose study in male and female patients with moderate to severe asthma in which patients will be stabilized on AEROVANT then doses of inhaled corticosteroids and LABA will be tapered. The hypothesis is that AEROVANT will improve asthma symptom control and decrease the need for inhaled corticosteroids and LABA, thus improving exacerbation incidence compared to placebo. Incidence of asthma exacerbation is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient, ≥ 18 years of age with a documented clinical history of asthma, has been treated for asthma and, in the opinion of the Investigator, is not fully controlled on current asthma therapy.
2. Patient satisfies, or has satisfied in the past, the GINA definition of moderate persistent to severe persistent asthma.
3. Patient has been maintained on moderate-to-high doses of ICS and LABA in the form of combination therapy or as individual agents (equivalent to fluticasone ≥ 250 mcg bid and salmeterol ≥ 50 mcg bid for ≥ 4 weeks before Screening [Visit 1]).
4. Patient has experienced an asthma exacerbation at least once in the past 2 years (defined here as use of physician prescribed oral corticosteroids or asthma requiring treatment increase approximately 4 times the baseline dose of inhaled corticosteroids or hospitalization due to asthma).
5. Patient has a pre-bronchodilator FEV1 ≥ 50% but ≤ 95% of the predicted value at both Screening (Visit 1) and Visit 2.
6. Patient demonstrates ≥ 12% reversibility (and a ≥ 200 mL difference) from prebronchodilator FEV1 within 15 to 30 minutes of receiving up to 4 puffs of a short-acting beta-agonist at Screening (Visit 1) or has ≥ 10% reversibility from pre-bronchodilator FEV1 plus a documented reversibility of ≥ 12% within the previous 12 months (documented methacholine or histamine sensitivity (PC20) <8mg/mL is also acceptable evidence or reversible airways disease).
7. Patient scores ≤ 20 on The Asthma Control Test™ at Screening (Visit 1) and Visit 2.
8. Female patient of childbearing potential or male patient and his female partner are practicing adequate and effective forms of contraception and agree to continue for the duration of the study. If female, must have a negative urine pregnancy test.
9. Patient has a pre-study medical history, physical examination, 12-Lead ECG, and safety laboratory test results within normal reference ranges or clinically acceptable to the Investigator.
10. Patient is a non-smoker for at least 6 months before Screening (Visit 1) and has a < 10 pack/year history of smoking.
11. Patient is medically stable for at least 8 weeks before Randomization (Visit 2), and the Investigator does not consider study participation to place the patient at increased risk of AEs (with the exception of possible asthma exacerbations).
12. Patient is able and willing to give written informed consent.

Exclusion Criteria:

1. Patient has a current diagnosis of respiratory disorder other than asthma (e.g., chronic bronchitis, bronchiectasis, emphysema, chronic obstructive pulmonary disease [COPD], etc).
2. Patient has received oral corticosteroid treatment within 8 weeks of Randomization (Visit 2)or patient has been intubated for ventilation in the past 5 years.
3. Patient has used any leukotriene antagonist within 1 week before Screening (Visit 1) or anti-IgE medications within 4 weeks of Screening (Visit 1).
4. Female patient is pregnant, breastfeeding, or not using an adequate method of contraception.
5. Patient has a clinically relevant medical history of very severs asthma that would preclude steroid reduction or sufficient compliance with the protocol.
6. Patient uses concomitant medications, including herbal, over-the-counter, or prescription medicines that, in the opinion of the Investigator, may affect the outcome of study endpoints and/or well-being of the patient.
7. Patient has a history of alcohol or substance abuse within 2 years of Screening (Visit 1).
8. Patient consumes more than 28 units (male) or 21 units (female) of alcohol a week (unit = 1 glass of wine = 1measure of spirits = ½ pint or 8 fluid ounces of beer).
9. Patient cannot communicate reliably with the Investigator or is unlikely to cooperate with the requirements of the study.
10. Patient has previously taken AEROVANT™ or another formulation of AER 001 (e.g., BAY 16-9996, pitrakinra).
11. Patient has participated in any clinical trial involving use of an investigational drug within 12 weeks of first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Incidence of exacerbation | 4 months

SECONDARY OUTCOMES:
In-clinic and daily pulmonary function | 4 months
Time to exacerbation after randomization | 4 months
Change from baseline in daily asthma symptom scores | 4 months
Change from baseline in daily beta-agonist reliever use | 4 months
Change from baseline in total IgE | 4 months
Change from baseline in fractional concentration of expired nitric oxide (FENO) | 4 months
Population pharmacokinetics | 4 months
General safety evaluation including lung function, blood pressure, heart rate, respiratory rate, temperature, ECG parameters, safety laboratory tests. | 4 months
SNP analysis for IL-4 and IL-13 relevant genes (Exploratory) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Sally Wenzel, M.D., Principal Investigator — University of Pittsburgh
Locations (71):
- United States (38):
  - Pulmonary Associates of Mobile, P.C., Mobile, Alabama
  - Allergy and Immunology Associates Ltd, Scottsdale, Arizona
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - Allergy Associates Medical Group Inc., San Diego, California
  - Institute of Healthcare Assessment Inc., San Diego, California
  - Allergy and Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - Allergy and Asthma Clinical Research Inc., Walnut Creek, California
  - Colorado Asthma and Allergy Research Centers, P.C., Centenniel, Colorado
  - Asthma and Allergy Associates P.C. and Research Center, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Florida Center for Asthma and Allergy Research, Miami, Florida
  - Allergy and Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - Partners in Asthma and Allergy Care, P.A., Valrico, Florida
  - Pulmonary Consultants of North Idaho, Coeur d'Alene, Idaho
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Allergy and Clinical Immunology, Bangor, Maine
  - The Brigham and Womens Hospital Inc., Boston, Massachusetts
  - North East Medical Research Associates, Inc, North Dartmouth, Massachusetts
  - Cardiopulmonary Associates of Missoula, Missoula, Montana
  - Pulmonary and Allergy Associates, Summit, New Jersey
  - ENT and Allergy Associates, Newburgh, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - IPS Research, Oklahoma City, Oklahoma
  - Allergy and Asthma Associates/Oak Street Medical P.C., Eugene, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Asthma and Allergy Research of New Jersey Inc., Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associates, PA, Upland, Pennsylvania
  - Asthma, Nasal Disease and Allergy Research Center of New England, Providence, Rhode Island
  - Greenville Pharmaceutical Research, Greenville, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Allergy and Asthma Research Center, P.A., San Antonio, Texas
  - Discovery Clinical Trials, LLC, San Antonio, Texas
  - Johnston Memorial Hospital, Abingdon, Virginia
- Hungary (11):
  - Dr. Kenessey Albert Kórház - Rendelőintézet, Balassagyarmat
  - Gyógyír XI Kht ( XI Kerületi Tüdőgondozó), Budapest
  - Margit Kórház, Csorna
  - Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkórháza, Deszk
  - Érd Városi Önkormányzat Szakorvosi Rendelőintézet, Érd
  - Szabolcs-Szatmár-Bereg Megyei Önkormányzat Jósa András Oktató Kórház, Nyíregyháza
  - Siofok Varos Korhaz-Rendelointezet, Siófok
  - Szarvasi Tüdőgyógyász Kft., Szarvas
  - Men For Care Kft. Százhalom Egészségügyi Központ, Százhalombatta
  - Vas Megyei Markusovszky Lajos Általános, Rehabilitációs és Gyógyfürdő Kórház, Szombathely
  - Komárom-Esztergom Megyei Önkormányzat Szent Borbála Kórháza, Tatabánya
- Poland (10):
  - Prywatny Gabinet Internistyczno - Alergologiczny, Bialystok
  - 10 Wojskowy Szpital Kliniczny z Poliklinika Kliniczny Oddzial Pulmonologiczny, Bydgoszcz
  - Specjalistyczny Zespol Chorob Pluc i Gruzlicy w Bystrej, Bystra
  - Medcare NZOZ, Gdansk
  - All-Med, Krakow
  - NZOZ Centrum Alergologii prof. Krzysztof Buczylko, Lodz
  - Poradnia Alergologii i Chorob Pluc SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im Norberta Barlicki, Lodz
  - AlergoTest SC, Lublin
  - NZOZ Centrum Medyczne Lucyna Andrzej Dymek, Strzelce Opolskie
  - Alergomed Specjalistyczna Przychodnia Lekarska sp zoo, Tarnów
- United Kingdom (12):
  - Barnsley District Hospital, Barnsley
  - Birmingham Heartlands Hospital, Birmingham
  - Queens Hospital, Burton-on-Trent
  - Woolpit Health Centre, Bury St Edmunds
  - Addenbrookes Hospital, Cambridge
  - Avondale Surgery, Chesterfield
  - Chesterfield Royal Hospital, Chesterfield
  - Colchester General Hospital, Colchester
  - Gartnavel General Hospital, Glasgow
  - Glenfield Hospital, Leicester
  - Hammersmith Hospital, London
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Slager RE, Otulana BA, Hawkins GA, Yen YP, Peters SP, Wenzel SE, Meyers DA, Bleecker ER. IL-4 receptor polymorphisms predict reduction in asthma exacerbations during response to an anti-IL-4 receptor alpha antagonist. J Allergy Clin Immunol. 2012 Aug;130(2):516-22.e4. doi: 10.1016/j.jaci.2012.03.030. Epub 2012 Apr 26. PMID 22541248